CLINICAL TRIAL: NCT06586034
Title: Culturally-Adapted Smoking Cessation Mobile App for Hispanic Individuals Who Smoke
Brief Title: Mobile Smoking Treatment for Hispanic Individuals Who Smoke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Michael J. Zvolensky, Ph.D., Hugh Roy and Lillie Cranz Cullen Distinguished University Professor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004990
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Smoking Cessation
Keywords: Mobile App; Smoking Cessation; Hispanic/Latino
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Impacto (Experimental): This is the mobile application to be developed and evaluated in this project.
  Interventions: Behavioral: Impacto (Mobile App)

INTERVENTIONS:
Behavioral: Impacto (Mobile App) — This is the mobile app to be developed and evaluated in this project. It is designed for both English and Spanish languages and is culturally tailored for Hispanic/Latino/Latinx individuals who smoke. Impacto will be developed for both iOS and Android platforms. The mobile app aims to aid smoking cessation by targeting elevated anxiety sensitivity.

SUMMARY:
The specific aims of the project are to develop and test a mobile application for smoking cessation for Hispanic individuals who smoke called Impacto.

DETAILED DESCRIPTION:
A total of 56 Hispanic individuals who smoke will be recruited for this project. Six (6) participants will complete usability/functionality testing of Impacto 2.0 in the English language for both iOS and Android. Following usability/functionality testing, a field test with 50 adult Hispanic individuals who smoke (50% English-speaking and 50% Spanish-speaking) will be recruited nationally and will receive Impacto 2.0 (50% Android and iOS platforms).

ELIGIBILITY:
Inclusion Criteria:

* 1) being Hispanic, 2) at least 18 years of age, 2) currently smoking (i.e., at least 5 cigarettes/day) biochemically verified by a CO > 7, 3), meeting criteria for high AS (cut-off score of 5 on the Short Scale Anxiety Sensitivity Index), 4) motivation to quit > 5 on a 10 pt. scale, 5) able to provide informed consent, 6) has daily access to their own iPhone or Android smartphone, and 7) is a fluent English or Spanish speaker.

Exclusion Criteria:

* 1) current participation in substance abuse treatment, 2) in psychotherapy for anxiety or depression, 3) concurrent use of medication for anxiety or depression, 4) active suicidality (ideation, intent, and/or plan), or 5) current psychosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
7-Day Point Prevalence Smoking Abstinence | End of treatment (Week 8)
  7-day point prevalence smoking status (verification via carbon monoxide).

SECONDARY OUTCOMES:
Anxiety Sensitivity | Baseline, week 4, and end of treatment (Week 8)
  Anxiety sensitivity will be assessed using the Short Scale Anxiety Sensitivity Index (SSASI).